CLINICAL TRIAL: NCT04060914
Title: LOwer Maintenance Dose TICagrelor in Acute Coronary Syndrome Patients Undergoing Percutaneous Coronary Intervention
Acronym: LOTIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Lin Yang, PHD, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZHEN HOSPITOL-LY-01
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Antiplatelet Therapy; Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: ticagrelor; clopidogrel; Percutaneous Coronary Intervention; Coronary Artery Disease; Adenosine
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ticagrelor(90mg) (Experimental)
  Interventions: Drug: Ticagrelor 90mg
- Ticagrelor(90/60mg) (Experimental)
  Interventions: Drug: Ticagrelor 90mg/60mg
- Clopidogrel(75mg) (Active Comparator)
  Interventions: Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — Ticagrelor 90 mg plus aspirin for 12 months
  Arms: Ticagrelor(90mg)
Drug: Ticagrelor 90mg/60mg — 1 month after treatment with ticagrelor 90 mg plus aspirin, followed by treatment with ticagrelor 60 mg plus aspirin for 11 months
  Arms: Ticagrelor(90/60mg)
Drug: Clopidogrel 75mg — Clopidogrel 75mg plus aspirin for 12 months
  Arms: Clopidogrel(75mg)

SUMMARY:
The hypothesis in this study was that ticagrelor switched to 60 mg after 1 month of standard dose, with antiplatelet activity that is not inferior to the standard dose and better than 75 mg clopidogrel for patients with ACS after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Agree to sign the Informed Consent;
* Male or female, ≥ 18 years of age, and ≤ 70 years of age
* Patient presents with acute coronary syndrome (ACS)
* Planned to undergo PCI
* Planned to DAPT for 1 year after PCI

Exclusion Criteria:

* Treatment with other investigational agents (including placebo) or devices within 30 days prior to randomization or planned use of investigational agents or devices prior to the Day 30 visit.
* Patients cannot use ticagrelor or clopidogrel due to contraindications or other reasons.
* Patients with active pathological hemorrhage or a history of intracranial hemorrhage
* Patient unable to receive 12 months of dual anti-platelet therapy
* Patient developing procedure-related complications such as stent thrombosis, coronary dissection, coronary perforation, cardiac tamponade or no-reflow during PCI
* Patient or physician refusal to enroll in the study
* History of intracranial hemorrhage
* Patient has a history of bleeding diathesis or coagulopathy
* Patient has an active pathological bleeding, such as active gastrointestinal (GI) bleeding
* Patient is pregnant, breastfeeding, or planning to become pregnant within 12 months
* Patient is receiving chronic oral anticoagulation therapy (i.e., vitamin K antagonist, direct thrombin inhibitor, Factor Xa inhibitor)
* Patient with cardiogenic shock or mechanical circulatory assist devices placed
* Patient with active liver diseases
* Patient with severe renal insufficiency (eGFR <30ml/min/1.73m2 based on simplified MDRD equation or CrCl <30ml/min based on Cockcroft-Gault equation)
* Patient has a malignancy or a life expectancy of less than one year
* Platelet count <100 000/μL, or hematocrit <32% or >52%, or white blood cell count <3000/μL
* Any other condition deemed by the investigator to place the patient at excessive risk of bleeding with ticagrelor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity index (PRI) | 90 days (±14)
  Platelet reactivity of ticagrelor or clopidogrel MD will be measured as PRI% using whole blood vasodilator-stimulated phosphoprotein (VASP) at 90 days after PCI.

SECONDARY OUTCOMES:
Occurrence of main adverse cardiovascular and cerebrovascular events (MACCE) | 1 year
  MACCE includes all-cause death, non-fatal stroke, non-fatal myocardial infarction (MI), and ischemic-driven revascularization.
The platelet aggregation ratio | 90 days (±14)
  Platelet aggregation of ticagrelor or clopidogrel MD will be measured using the Light Transmittance Aggregometry method at day 90 after PCI.
Plasma adenosine concentration | 90 days (±14)
  Plasma adenosine concentration in the three treatment groups will be measured using the HPLC-MS at day 90 after PCI.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided